CLINICAL TRIAL: NCT04515745
Title: The Effects of an Intensive Lifestyle Intervention for Type 2 Diabetes on Disability Insurance Applications, Receipt, and Payments
Brief Title: The Effects of an Intensive Lifestyle Intervention for Type 2 Diabetes on Disability Insurance
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Southern California (Other); Wake Forest University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: UP-16-00706-2; 5R01DK107552 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ILI/Treatment group: This group includes Look AHEAD participants who were initially assigned to the intensive lifestyle intervention (ILI), consented to administrative data linkages, and were successfully linked to Social Security Administration (SSA) databases.
  Interventions: Behavioral: Intensive lifestyle intervention (ILI)
- DSE/Control group: This group includes Look AHEAD participants who were initially assigned to the diabetes support and education (DSE) control arm, consented to administrative data linkages, and were successfully linked to SSA databases.
  Interventions: Behavioral: Diabetes support and education (DSE)

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention (ILI) — Lifestyle intervention focused on weight loss through diet and physical activity
  Groups: ILI/Treatment group
Behavioral: Diabetes support and education (DSE) — Behavioral intervention focused on diabetes support and education
  Groups: DSE/Control group

SUMMARY:
Starting in 2001, the Look AHEAD study randomized patients with type 2 diabetes to an intensive lifestyle intervention (ILI) focused on weight loss versus a control group receiving diabetes education ("Diabetes Support and Education"). The ILI successfully reduced weight, improved diabetes control, and functional status, among other outcomes. In this study, the investigators will compare participation in federal disability insurance programs between the ILI and the control group during and after the intervention period (2001-2017).

DETAILED DESCRIPTION:
Starting in 2001, the Look AHEAD study randomized 5145 patients with type 2 diabetes to an intensive lifestyle intervention (ILI) focused on weight loss versus a control group receiving diabetes education ("Diabetes Support and Education").The Look AHEAD study tested whether participants with type 2 diabetes assigned to an intensive lifestyle intervention (ILI) for weight loss exhibited reductions in cardiovascular morbidity and mortality, relative to a control group receiving usual care and diabetes support and education. During the 12-year intervention period, the ILI led to persistent reductions in weight, waist circumference, and hemoglobin A1c and improvements in physical fitness, among other clinical benefits. After the conclusion of the intervention in 2012, participants were consented to be linked with administrative data. The investigators attempted to link 3188 consenting participants with Social Security Administration databases. Of these, the investigators were able to successfully link 3093 participants. In this study, the investigators will compare participation in federal disability insurance programs including Social Security Disability Insurance (SSDI) and disability-related Supplemental Security Income (SSI) between the linked ILI and the control group during and after the intervention period (2001-2017). The investigators will investigate ILI-versus-control differences in whether participants ever applied or received benefits from SSDI and SSI. The investigators will also investigate ILI-versus-control differences in applications and benefit receipt in each year after randomization, relative to a pre-randomization assessment period. The investigators will use both multivariate regression controlling for baseline participant characteristics and clinic site and also survival analyses that estimate whether the time until SSDI or SSI application or benefit receipt differs between the ILI and control groups.

ELIGIBILITY:
(Note: age limits above are at time of randomization, which occurred between 2001-2004)

Inclusion Criteria:

* Look AHEAD participation: met age requirements and other criteria at time of study enrollment which occurred between 2001-2004 (as noted in Look AHEAD Research Group (2013))
* Consented to administrative data linkages
* Provided individual identifiers that could be linked with SSA databases
* Were successfully linked to SSA data

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes Look AHEAD participants that consented to administrative data linkages, provided individual identifiers that could be linked with SSA data, and were successfully linked to SSA data.
Sampling Method: Non-Probability Sample
Enrollment: 3091 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Ever received public disability program benefits (Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI)) | This measure will capture program participation between randomization (randomization occurred between 2001-2004) through 2017
  This is based on Social Security Administration data on SSDI and SSI benefits, SSDI entitlement and SSI eligibility.
Ever applied for public disability program benefits (Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI)) | From initial randomization (randomization occurred between 2001-2004) through 2017
  This is based on Social Security Administration data on applications for SSDI and SSI.

SECONDARY OUTCOMES:
Ever received Social Security Disability Insurance (SSDI) benefits | This measure will capture program participation occurring between randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data indicating SSDI benefits and SSDI entitlement.
Ever received disability-related Supplemental Security Income (SSI) benefits | This measure will capture program participation occurring between randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data indicating SSI benefits and SSI eligibility.
Ever applied for Social Security Disability Insurance (SSDI) benefits | From initial randomization (occurred between 2001-2004) through 2017
  This measure is based on Social Security Administration data on applications for SSDI.
Ever applied for disability-related Supplemental Security Income (SSI) benefits | From initial randomization (occurred between 2001-2004) through 2017
  This measure is based on Social Security Administration data on applications for SSI.
Total person-months of Social Security Disability Insurance (SSDI) benefits received | From initial randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data on SSDI and SSDI entitlement.
Total person-months of disability-related Supplemental Security Income (SSI) benefits received | From initial randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data on SSI benefits and SSI eligibility.
Total person-months of Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits received | From initial randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data on SSDI and SSI benefits, SSDI entitlement and SSI eligibility.
Total Social Security Disability Insurance (SSDI) payments | From initial randomization (occurred between 2001-2004) through 2017.
  This is based on Social Security Administration data on SSDI payments, adjusting for inflation.
Total disability-related Supplemental Security Income (SSI) payments | From initial randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data on SSI payments, adjusting for inflation.
Total disability payments (Social Security Disability Insurance (SSDI) and disability-related Supplemental Security Income (SSI)) | From initial randomization (occurred between 2001-2004) through 2017
  This based on Social Security Administration data on SSDI and SSI payments, adjusted for inflation.
Received Social Security Disability Insurance (SSDI) benefits | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data indicating SSDI benefits and SSDI entitlement.
Received disability-related Supplemental Security Income (SSI) benefits | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data indicating SSI benefits and SSI eligibility.
Received Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on SSDI and SSI benefits, SSDI entitlement and SSI eligibility.
Application for Social Security Disability Insurance (SSDI) benefits | 12-month intervals relative to randomization occurring between 2001-2017.
  This measure is based on Social Security Administration data on applications for SSDI.
Application for disability-related Supplemental Security Income (SSI) benefits | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on applications for SSI.
Application for Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits. | 12-month intervals relative to randomization occurring between 2001-2017
  This measure is based on Social Security Administration data on applications for SSDI and SSI.

OTHER OUTCOMES:
Ever received disability benefits (Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits) within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data on SSDI and SSI benefits, SSDI entitlement and SSI eligibility.
Ever received Social Security Disability Insurance (SSDI) benefits within 8 years of randomization | This measure will capture program participation within 8 years of randomization (occurred 2001-2004)
  This is based on Social Security Administration data indicating SSDI benefits received and SSDI entitlement.
Ever received disability-related Supplemental Security Income (SSI) benefits within 8 years of randomization | This measure will capture program participation within 8 years of randomization (occurred 2001-2004)
  This is based on Social Security Administration data indicating SSI benefits received and SSI eligibility.
Ever applied for disability benefits (Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data indicating applications for SSDI or SSI.
Ever applied for Social Security Disability Insurance (SSDI) benefits within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data indicating applications for SSDI.
Ever applied for disability-related Supplemental Security Income (SSI) benefits within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data indicating applications for SSI.
Total person-months of Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits received within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data on SSDI and SSI benefits, SSDI entitlement and SSI eligibility.
Total person-months of Social Security Disability Insurance (SSDI) benefits received within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data on SSDI and SSDI entitlement.
Total person-months of disability-related Supplemental Security Income (SSI) benefits received within 8 years of randomization | The first 8 years following randomization, which occurred from 2001 to 2004.
  This is based on Social Security Administration data on SSI benefits and SSI eligibility.
Person-months of Social Security Disability Insurance (SSDI) benefits received | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on SSDI and SSDI entitlement.
Person-months of disability-related Supplemental Security Income (SSI) benefits received | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on SSI and SSI eligibility.
Person-months of Social Security Disability Insurance (SSDI) or disability-related Supplemental Security Income (SSI) benefits received | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on SSDI and SSI benefits, SSDI entitlement and SSI eligibility.
Social Security Disability Insurance (SSDI) payments | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on SSDI payments, adjusting for inflation.
Disability-related Supplemental Security Income (SSI) payments | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data on SSI payments, adjusting for inflation.
Disability payments (Social Security Disability Insurance (SSDI) and disability-related Supplemental Security Income (SSI)) | 12-month intervals relative to randomization occurring between 2001-2017
  This based on Social Security Administration data on SSDI and SSI payments, adjusted for inflation.
Labor force participation conditional on enrollment in disability programs | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data indicating labor force participation among recipients of Social Security Disability Insurance and Supplemental Security Income.
Annual labor market earnings conditional on enrollment in disability programs | 12-month intervals relative to randomization occurring between 2001-2017
  This is based on Social Security Administration data indicating earnings among recipients of Social Security Disability Insurance and Supplemental Security Income.
Ever participated in labor force conditional on enrollment in disability programs. | From initial randomization (occurred between 2001-2004) through 2017
  This is based on Social Security Administration data indicating labor force participation while individuals received Social Security Disability Insurance or Supplemental Security Income benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Huckfeldt, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No
Use of Social Security Administration data is restricted under a data use agreement between the Social Security Administration and Wake Forest.

REFERENCES:
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131